CLINICAL TRIAL: NCT00154570
Title: Integrating Simultaneous Recording of 24 Hour Esophageal pH and Electrogastrography to Investigate the Mechanism of Reflux Esophagitis
Brief Title: 24 Hour Esophageal and Electrogastrography to Investigate the Mechanism of Reflux Esophagitis
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: National Taiwan University Hospital (Other)
Other Study IDs: 9261701469
Record Dates: First submitted 2005-09-09; First posted 2005-09-12 (Estimated); Last update posted 2005-11-22 (Estimated); Status verified 2004-02

CONDITIONS: Reflux Esophagitis
Keywords: reflux esophagitis; 24 hour esophageal pH; electrogastrography (EGG); Running Spectral Analysis (RSA)
MeSH Terms: conditions — Esophagitis, Peptic

STUDY DESIGN:
Observational Model: Defined Population | Time Perspective: Other

INTERVENTIONS:
Device: EGG, 24 hour esophageal pH monitor

SUMMARY:
We hypothesize that gastric dysrhythmias may predispose the occurrence of gastroesophageal reflux.

DETAILED DESCRIPTION:
Gastroesophageal regurgitation with acid is considered the main cause of reflux esophagitis, but the current theory of transient relaxation of LES (TLESR) fails to explain all the mechanisms of reflux esophagitis, for a rather high proportion of reflux esophagitis patients has concomitant other functional gastrointestinal disorder, particularly gastric motility dysfunction. Thus, these patients could even not effectively respond to proton pump inhibitor alone. Abnormal gastric emptying and antral dysmotility has been considered related to reflux esophagitis. EGG is a promising noninvasive tool in study of gastric electric activity and motility, and the application of gastric electric stimulation (GES) in the modulation of gastric motility disorder and even reflux esophagitis has been in proceeding; however, there is lacking study by using EGG to integrate gastric electrical potentials, gastric motility and gastroesophageal reflux in investigating the mechanism of reflux esophagitis till now; especially, no known literature by combined simultaneous prolong ambulatory esophageal pH and EGG recordings has been reported. It has been known in EGG study that gastric dysrhythmias (tachy- and brady-) related smooth muscle function of stomach and dysfunctional gastric emptying.

In a preliminary findings of simultaneous prolong ambulatory esophageal pH and EGG recordings by our study group, we found that gastroesophageal reflux with acid tends in the status of abnormal RSA. Thus, we propose the following hypotheses: (1) Gastric dysrhythmias may predispose the occurrence of gastroesophageal reflux. We plan to use the recorder of esophageal pH and gastric electric potentials developed in Institute of Medical Engineering, National Taiwan University, combining with the unique design of simultaneous 24 hour ambulatory esophageal pH and EGG recordings and Matlab analysis of RSA-pH, to explore the relationship of gastric electric potentials and reflux esophagitis.

Objectives: (1) Use simultaneous 24 hour ambulatory esophageal pH metry and EGG to integrate RSA and esophageal pH to explore whether a specific RSA prone to gastroesophageal reflux; or whether gastroesophageal reflux influence gastric electric activity; (2) Integrate RSA and esophageal pH with event of GI symptoms and daily activity to explore whether symptoms are resulted from acid reflux or gastric dysrhythmias.

Materials and methods: Recruits 25 healthy and 25 previously diagnosed reflux esophagitis patients as volunteers to receive the followings:

1. GI and GERD symptom questionnaire with score of severity and frequency, and quality of life (QoL).
2. 24-hour ambulatory esophageal pH recording: total numbers of reflux episodes, total duration of pH < 4 and DeMester score. They will be classified into: pathologic (pH < 4, > 4%且DeMeester score > 14.72 ) and non-pathologic (pH < 4, < 4% and DeMeester score < 14.72).
3. 24-hour ambulatory EGG recording: Use RSA to evaluate the quantity and quality of gastric electrical potentials. They will be classified into normal (3cpm), tachyrhythmia (> 3cpm), and bradyrhythmia (< 3cpm) three groups.
4. Use Matlab soft ware to integrate the data of simultaneous 24-hour esophageal pH value and RSA with events of symptoms and daily activities (meal time, postprandial, fasting, sleeping, and exercise).

ELIGIBILITY:
Inclusion Criteria:

* GERD questionnaire with heartburn or acid regurgitation with a frequency at least once weekly.
* Endoscopic esophagitis.

Exclusion Criteria:

* A history of esophageal, gastric or abdominal surgery.
* Gastric or esophageal cancer.
* Esophageal varices.
* Concomittant severe systemic disease.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50
Dates: Start 2004-02; Study Completion 2005-08

CONTACTS AND LOCATIONS:
Overall Officials: Bor-Ru Lin, M.D., Principal Investigator — National Taiwan University Hospital
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan